CLINICAL TRIAL: NCT05562336
Title: Optical Coherence Tomography Angiography Criteria Of The Choroidal Neovascular Membrane In Wet Age Related Macular Degeneration And In Pathological Myopia (Comparative Study).
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Arwa Mostafa Ahmed, Principal investigator, Sohag University
Other Study IDs: Soh-Med-22-09-03
Record Dates: First submitted 2022-09-22; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Choroidal Neovascular Membrane In Wet Age Related Macular Degeneration And In Pathological Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with age related macular degeneration with CNV
  Interventions: Device: Optical coherence tomography angiography
- Patients with pathological myopia with CNV
  Interventions: Device: Optical coherence tomography angiography

INTERVENTIONS:
Device: Optical coherence tomography angiography — Optical coherence tomography (OCT) is a noninvasive imaging method that uses reflected light to create pictures of the back of your eye

SUMMARY:
This study aims to compare choroidal neo-vascular membrane criteria in cases of age-related macular degeneration and cases of pathological myopia.

DETAILED DESCRIPTION:
All patients will be examined by optical coherence tomography (OCT) and optical coherence tomography angiography (OCT-angio) .

The size, the location, the criteria of the choriodal neovascular membrane will be examined and imaged.

Study include 50 cases of CNV in age related macular degeneration and 50 cases of CNV in pathological myopia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age related macular degeneration should be at least 50 years of age with CNV with no other causes.

Patients with pathological myopia where axial length more than 26 mm or refractive power more than -6 diopter with CNV in OCT with clear media and OCT-angio can be used.

Exclusion Criteria:

* Exclude other pathological causes of CNV .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cnv in age related macular degeneration and in pathological myopia
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
choroidal neo-vascular membrane criteria in cases of age-related macular degeneration and cases of pathological myopia | through study completion, an average of 1 year
  choroidal neo-vascular membrane identified by Optical Coherence Tomography Angiography

REFERENCES:
- [Background] Hee MR, Baumal CR, Puliafito CA, Duker JS, Reichel E, Wilkins JR, Coker JG, Schuman JS, Swanson EA, Fujimoto JG. Optical coherence tomography of age-related macular degeneration and choroidal neovascularization. Ophthalmology. 1996 Aug;103(8):1260-70. doi: 10.1016/s0161-6420(96)30512-5. PMID 8764797
- [Background] Secretan M, Kuhn D, Soubrane G, Coscas G. Long-term visual outcome of choroidal neovascularization in pathologic myopia: natural history and laser treatment. Eur J Ophthalmol. 1997 Oct-Dec;7(4):307-16. doi: 10.1177/112067219700700401. PMID 9457451
- [Background] Miller DG, Singerman LJ. Vision loss in younger patients: a review of choroidal neovascularization. Optom Vis Sci. 2006 May;83(5):316-25. doi: 10.1097/01.opx.0000216019.88256.eb. PMID 16699445
- [Background] Kovach JL, Schwartz SG, Flynn HW Jr, Scott IU. Anti-VEGF Treatment Strategies for Wet AMD. J Ophthalmol. 2012;2012:786870. doi: 10.1155/2012/786870. Epub 2012 Feb 28. PMID 22523653